CLINICAL TRIAL: NCT07386717
Title: Upadacitinib Versus IL-17 Inhibitors in Patients With Psoriatic Arthritis: A Cohort Study
Brief Title: Upadacitinib Versus IL-17 Inhibitors in Patients With Psoriatic Arthritis
Acronym: UVIPWP
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UVIPWP_V1
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis; Upadacitinib; Interleukin-17 Inhibitors
Keywords: Interleukin-17 Inhibitors; Upadacitinib; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Upadacitinib-Treated PsA Patients: Adult patients with psoriatic arthritis receiving upadacitinib as part of routine clinical care and followed for 24 weeks.
- Cohort 2: IL-17 Inhibitor-Treated PsA Patients: Adult patients with psoriatic arthritis receiving interleukin-17 inhibitors (e.g., secukinumab or ixekizumab) as part of routine clinical care and followed for 24 weeks.

SUMMARY:
Psoriatic arthritis (PsA) is a chronic inflammatory disease with heterogeneous musculoskeletal and dermatologic manifestations, leading to significant functional impairment and reduced quality of life. Although targeted therapies such as Janus kinase inhibitors and interleukin-17 inhibitors have demonstrated efficacy in randomized controlled trials, real-world comparative evidence between these treatment strategies remains limited.

This observational cohort study aims to compare the real-world effectiveness and safety of upadacitinib and interleukin-17 inhibitors in patients with PsA over a 24-week follow-up period. By evaluating clinical outcomes under routine clinical practice conditions, this study seeks to provide evidence to support individualized treatment selection in PsA management.

DETAILED DESCRIPTION:
This is a real-world, observational cohort study conducted at Peking University First Hospital. Adult patients diagnosed with psoriatic arthritis will be enrolled and followed for 24 weeks in routine clinical practice.

Participants will be categorized into two cohorts based on treatment exposure at baseline: patients receiving upadacitinib and patients receiving interleukin-17 inhibitors. Treatment decisions are made by treating physicians according to standard clinical practice and are not influenced by the study protocol.

Clinical assessments will be performed at baseline and during routine follow-up visits within the 24-week observation period. Effectiveness outcomes will be evaluated across musculoskeletal and dermatologic domains, and safety outcomes will be monitored throughout follow-up. This study does not involve experimental interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of psoriatic arthritis according to established classification criteria
* Treatment with upadacitinib or an interleukin-17 inhibitor at baseline
* Availability of baseline and follow-up clinical data over 24 weeks

Exclusion Criteria:

* Diagnosis of other inflammatory arthritides
* History of malignancy or severe uncontrolled infection
* Incomplete clinical data preventing outcome assessment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of psoriatic arthritis according to established classification criteria
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness of treatment | Baseline to Week 24
  Changes in joint and skin disease activity assessed using validated clinical measures during the 24-week follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided